CLINICAL TRIAL: NCT01483300
Title: Effectiveness and Toxicity of Gemcitabine/Lobaplatin Versus Gemcitabine/Cisplatin as Second-line Treatment in Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Qingyuan Zhang, Vice president of Cancer Hospital of Harbin Medical University, Harbin Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BC001
Record Dates: First submitted 2011-11-25; First posted 2011-12-01 (Estimated); Last update posted 2012-01-24 (Estimated); Status verified 2012-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; gemcitabine; lobaplatin; cisplatin
MeSH Terms: conditions — Breast Neoplasms | interventions — lobaplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lobaplatin (Experimental): gemcitabine plus lobaplatin
  Interventions: Drug: lobaplatin
- cisplatin (Active Comparator): gemcitabine plus cisplatin
  Interventions: Drug: cisplatin

INTERVENTIONS:
Drug: lobaplatin — Gemcitabine 1000 mg/m2 d1, 8; Lobaplatin 30mg/m2 d1 q 3 weeks
  Arms: lobaplatin
Drug: cisplatin — Gemcitabine 1000 mg/m2 d1, 8; Cisplatin 25 mg/m2 d1-3 q 3 weeks
  Arms: cisplatin

SUMMARY:
Gemcitabine plus cisplatin has been proved to be an effective regimen as second-line treatment for metastatic breast cancer patients, especially for those previously treated with anthracyclines and taxanes. Lobaplatin, as the third generation of new cancer drug platinum, has a similar anticancer activity to cisplatin, but less kidney toxicity and gastrointestinal reaction. The purpose of the study is to compare the efficacy and safety of gemcitabine/lobaplatin versus gemcitabine/cisplatin in patients with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic breast cancer
* Disease progression during or after previous 1st line chemotherapy
* Scheduled to receive 2nd line chemotherapy.
* Measurable disease, defined as a least one lesion that can be accurately measured in at least one dimension
* 18 years of age or older
* ECOG performance status of 0-2
* Life expectancy of greater than 6 months

Exclusion Criteria:

* Previous treatment with one of the study drugs
* Application of other cytotoxic chemotherapy or radiotherapy
* Insufficent renal function (creatinine clearance < 60ml/min)
* Clinically unstable brain metastasis
* Pregancy or lactation
* History of other malignancy within last 5 years.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-11; Primary Completion 2014-08 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 4 weeks after chemotherapy
  Overall response rate (ORR) defined as complete response(CR) + partial response(PR) + stable disease (SD)

SECONDARY OUTCOMES:
Time to progression | one year after last patient in
  Time to progression defined as time from randomization to disease progress.
Overall Survival | one year after last patient in
  Overall survival defined as time from randomization to death from any cause.
Treatment related toxicity | 4 weeks after chemotherapy
  Treatment related toxicities will be recorded as chemotherapy toxicity grades in hematologic, renal, hepatic and gastrointestinal system.

CONTACTS AND LOCATIONS:
Overall Officials: Qingyuan Zhang, MD, Study Director — Cancer Hospital of Harbin Medical University; Xinmei Kang, MD, Principal Investigator — Cancer Hospital of Harbin Medical University
Locations (1):
- Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang, China